CLINICAL TRIAL: NCT06978855
Title: Efficacy of Wrist Acupressure Band on Sleep Quality in Medical Trainees: A Single-Blinded Cross-Over Randomized Clinical Trial
Brief Title: Efficacy of Wrist Acupressure Band on Sleep Quality in Medical Trainees
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Georges Assaf, Clinical Assistant Professor of Family Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: SBS-2024-0323
Record Dates: First submitted 2025-05-16; First posted 2025-05-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sleep; SLEEP DISTURBANCES Nec in ICD9CM; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): this group will be assigned to apply the wrist band at the intervention acupressure point studied
  Interventions: Device: Wrist band acupressure application to P6 point
- control (Sham Comparator): this group will be assigned to apply the wrist band to a sham point
  Interventions: Device: Wrist band acupressure application to sham point

INTERVENTIONS:
Device: Wrist band acupressure application to P6 point — The intervention group received standardized instructions for applying the wristband to the P6 acupressure point on their wrist, with daily application scheduled from 8 pm to 8 am. Those who have night shifts will be asked to apply the wrist band for 12 hours after the end of their shift the intervention was applied for 30 days.
  At the end of the first phase the participants will be asked to avoid applying the wrist band for 7 days, to allow a washout period before crossing over.
  Arms: intervention
Device: Wrist band acupressure application to sham point — the control group will receive standardized instructions to apply the wristband to a sham point, with daily application from 8 pm to 8 am. Those who have night shifts will be asked to apply the wrist band for 12 hours after the end of their shift. This will occur for 30 days. At the end of the first phase the participants will be asked to avoid applying the wrist band for 7 days, to allow a washout period before crossing over.
  Arms: control

SUMMARY:
Background: Medical trainees frequently experience sleep disturbances, with shift work being a major contributing factor impacting their performance and overall wellbeing. Traditional treatments for sleep disorders often involve medications and hypnotics with potential side effects, highlighting the need for alternative strategies. Acupressure, particularly at the P6 (Neiguan) point, has shown promise in improving sleep and reducing anxiety.

Objective: This study aimed to evaluate the efficacy of wristband acupressure applied to the P6 point in improving sleep quality, anxiety levels, and overall well-being among medical trainees.

Methods: A single-blinded, cross-over randomized controlled trial was conducted at the American University of Beirut Medical Center (AUBMC), involving 10 medical trainees. Participants were randomized in blocks to either the intervention group, receiving wristband acupressure at the P6 point, or the control group, receiving acupressure at a sham point. Standardized, validated questionnaires were used to assess sleep quality (PSQI), anxiety (GAD-7), and well-being (WHO-5) before and after each intervention period. Ethical approval was obtained from the Institutional Review Board, and participant confidentiality was maintained

ELIGIBILITY:
Inclusion Criteria:

Residents, Fellows and Med-4 students at AUB.

Exclusion Criteria:

* Being enrolled in another sleep study
* Currently on Sleep Medications: Benzodiazepines, antihistamines, muscle relaxants, magnesium supplements, herbal supplements that help with sleep including Chamomile, Ashwaghanda and Melatonin
* Daily alcohol consumers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 1 month
  Pittsburgh Sleep Quality Index (PSQI) score, ranging from 0 to 21. Higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | 1 month
  Generalized Anxiety Disorder-7 (GAD-7): Scores range from 0 to 21, with higher scores indicating greater severity of anxiety symptoms.
World Health Organization Well-Being Index (WHO-5) | 1 month
  World Health Organization Well-Being Index (WHO-5): Raw scores range from 0 to 25 and are multiplied by 4 to give a percentage score from 0 to 100. Higher scores indicate better well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- American university of Beirut, Beirut, Beyrouth, Lebanon